CLINICAL TRIAL: NCT00223704
Title: Bradykinin Receptor Antagonism During Cardiopulmonary Bypass
Acronym: BRAC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Mias Pretorius, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB #051171; HL085740-02
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Cardiopulmonary Bypass; Inflammation; Fibrinolysis; Surgery
Keywords: Coronary Artery Bypass; Blood Transfusion; Bradykinin Receptor Antagonism; Anti-Inflammatory Agents; Antifibrinolytic Agents
MeSH Terms: conditions — Inflammation | interventions — icatibant; Aminocaproic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HOE 140 (Experimental): Bradykinin receptor antagonist
  Interventions: Drug: HOE 140
- Aminocaproic Acid (Active Comparator): Antifibrinolytic
  Interventions: Drug: Aminocaproic Acid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HOE 140 — HOE 140 (a bradykinin B2 receptor antagonist) was started in the operating room after induction of anesthesia and before heparinization, continued throughout the bypass period, and discontinued at the end of surgery. HOE 140 was given as an intravenous bolus of 22 µg/kg over one-half hour followed by an infusion of 18 µg/kg/hr.
  Other Names: Icatibant
  Arms: HOE 140
Drug: Aminocaproic Acid — Aminocaproic acid (an antifibrinolytic drug) was started in the operating room after induction of anesthesia and before heparinization, continued throughout the bypass period, and discontinued at the end of surgery. Aminocaproic acid was given as an intravenous bolus of 100 mg/kg over one-half hour followed by an infusion of 30 mg/kg/hr.
  Other Names: Amicar; EACA
  Arms: Aminocaproic Acid
Drug: Placebo — Normal saline (placebo) was started in the operating room after induction of anesthesia and before heparinization, continued throughout the bypass period, and discontinued at the end of surgery.
  Other Names: Placebo/Normal Saline
  Arms: Placebo

SUMMARY:
Each year over a million patients worldwide undergo cardiac surgery requiring cardiopulmonary bypass (CPB). CPB is associated with significant morbidity including the transfusion of allogenic blood products, inflammation and hemodynamic instability. In fact, approximately 20% of all blood products transfused are associated with coronary artery bypass grafting procedures. Transfusion of allogenic blood products is associated with well-documented morbidity and increased mortality after cardiac surgery. Enhanced fibrinolysis contributes to increased blood product transfusion in the perioperative period. The current proposal tests the central hypothesis that endogenous bradykinin contributes to the hemodynamic, fibrinolytic and inflammatory response to CPB and that bradykinin receptor antagonism will reduce hypotension, inflammation and transfusion requirements. In SPECIFIC AIM 1 we will test the hypothesis that the fibrinolytic and inflammatory response to CPB differ during ACE inhibition and angiotensin II type 1 receptor antagonism. In SPECIFIC AIM 2 we will test the hypothesis that bradykinin B2 receptor antagonism attenuates the hemodynamic, fibrinolytic, and inflammatory response to CPB. In SPECIFIC AIM 3 we will test the hypothesis that bradykinin B2 receptor antagonism reduces the risk of allogenic blood product transfusion in patients undergoing CPB. These studies promise to provide important information regarding the effects of drugs that interrupt the RAS and generate new strategies to reduce morbidity in patients undergoing CPB.

DETAILED DESCRIPTION:
Morbidity of cardiopulmonary bypass. Each year more than a million patients worldwide undergo cardiac surgery. Nearly all cardiac surgeries are performed on unbeating hearts supported by CPB. Although the use of off-pump coronary artery bypass surgery procedures are increasing, concerns regarding incomplete revascularization and reduced venous graft patency limit the use of this technique to specific patients. CPB activates various humoral cascades including the coagulation cascade, the KKS, the fibrinolytic cascade, and causes a systemic inflammatory response syndrome. Activation of these systems can lead to hypotension, fever, disseminated intravascular coagulation, diffuse tissue edema, or, in extreme cases, to multiple organ failure. Activation of the KKS contributes to the hemodynamic perturbations, fibrinolysis and inflammatory response observed in patients undergoing CPB. Aprotinin, a non-specific serine protease inhibitor, that works in part by decreasing bradykinin generation, decreases fibrinolysis, hypotension and the systemic inflammatory response associated with CPB. Aprotinin decreases blood loss and transfusion requirements, however, its use is mainly limited to redo-cardiac surgery because of cost. Other factors that may limit the widespread use of aprotinin include an increased risk for renal dysfunction, allergic reaction and non-specificity of the drug. Bradykinin mediates most of the effects of the KKS. Thus, bradykinin receptor antagonism has the potential to modulate the effects of KKS activation during CPB. The purpose of this proposal is to test the hypothesis that endogenous bradykinin contributes to the hemodynamic, fibrinolytic and inflammatory response to CPB and that bradykinin receptor antagonism will reduce hypotension, inflammation and transfusion requirements. The proposed studies promise to lead to novel therapies to reduce morbidity associated with CPB.

Cardiopulmonary bypass activates the kallikrein-kinin system (KKS). Several groups, including ours, have reported that bradykinin concentrations increase during CPB. For example, Campbell et al demonstrated that bradykinin levels increase 10 to 20-fold during the first 10 minutes of CPB, returned to basal levels by 70 minutes of CPB and remained 1.7 to 5.2-fold elevated after CPB. Plasma and tissue kallikrein were reduced by 80 and 60% respectively, during the first minute of CPB. Similarly, we have demonstrated that bradykinin increases significantly during CPB and that ACE inhibition and smoking potentiate the kinin response during CPB.

Fibrinolytic response to cardiopulmonary bypass. CPB increases t-PA antigen and activity in a time-dependent manner. The fibrinolytic response during CPB is heterogeneous, with t-PA levels varying as much as 250-fold. The mechanism of t-PA release during CPB is likely multifactorial. As outlined above, we and others have shown that CPB increases bradykinin, a potent stimulus to t-PA release. In addition, thrombin or complement generated during CPB may stimulate the release of t-PA from endothelium. In addition to the changes in t-PA concentrations during CPB, PAI-1 activity falls because of hemodilution and the rise in t-PA release which consumes active PAI-1. Plasmin generation increases over 100-fold while D-dimer generation increases 200-fold within 5 minutes of CPB initiation. For the remainder of the CPB, average plasmin and D-dimer levels remain 20-fold to 30-fold above baseline levels. The postoperative period is marked by a systemic inflammatory response caused by a combination of CPB and surgery producing an acute -phase response that results in increased PAI-1 production. PAI-1 levels begin to rise about 2 hours after surgery. Once CPB is over, PAI-1 levels continue to rise and peak during the first 12-36 hours postoperatively and return to normal by the second postoperative day. Thus, the fibrinolytic response to CPB is characterized by an initial hyperfibrinolytic phase that begins with a rapid rise in t-PA, plasmin, and D-dimer concentrations followed by a postoperative hypofibrinolytic phase associated with a rise in PAI-1 secretion and a fall in t-PA concentrations.

Interaction between the renin-angiotensin system (RAS), the KKS and fibrinolytic system. There is evidence that fibrinolytic balance is regulated by the RAS and the KKS. ACE is strategically poised to control fibrinolytic balance by promoting the breakdown of bradykinin and the conversion of Ang I to Ang II. Ang II causes the release of PAI-1 thus inhibiting fibrinolysis. Bradykinin stimulates t-PA release through its B2 receptor. ACE inhibition decreases PAI-1 antigen levels and increases endothelial t-PA release through endogenous bradykinin. In addition, ACE inhibition enhances exogenous bradykinin-mediated vasodilation and t-PA release. The augmentation of bradykinin-induced vasodilation, the increase in t-PA and the decrease in PAI-1 described with ACE inhibition in patients with ischemic heart disease may contribute to the primary mechanism of the anti-ischemic effects associated with chronic ACE inhibitor therapy. We have demonstrated that inpatients undergoing coronary artery bypass grafting (CABG) requiring CPB, not only did ACE inhibition increase fibrinolytic activity by decreasing PAI-1 antigen and increasing t-PA activity, but also enhanced the kinin response. Increased PAI-1 concentrations in the perioperative period are associated with acute vein graft thrombosis. Thus, ACE inhibitors have a potential to reduce the risk of acute graft thrombosis through their effects on Ang II generation by attenuating the PAI-1 response after CABG. As opposed to the beneficial effects of ACE inhibition on PAI-1, the augmentation of the kinin response during CPB may have detrimental effects including increased fibrinolysis with consequent bleeding and hypotension. The effect of angiotensin II type 1 (AT1) receptor antagonist on the fibrinolytic response to CPB is not known. Inpatients with essential hypertension AT1 receptor antagonist decreases PAI-1 antigen in some but not other studies. In Specific Aim 1 we will test the hypothesis that angiotensin-converting enzyme inhibitors and AT1 receptor antagonist modulate the fibrinolytic and inflammatory response to CPB differently.

Bradykinin receptor antagonism could reduce the hypotensive response to CPB. Low systemic vascular resistance (SVR) commonly occurs during and early after CPB. It is usually transient and easy to treat. Occasionally, patients have a more severe and persistent fall in SVR, referred to postoperative vasodilatory shock. Risk factors for vasodilatory shock includes the preoperative use of ACE inhibitors, low left ventricular ejection fraction and heart failure syndrome. Treatment is frequently required to maintain adequate perfusion pressure during CPB and to establish satisfactory hemodynamics when ready to separate the patient from bypass. This usually entails counteracting the effect of the vasodilatory mediators by administration of drugs such as norepinephrine or phenylephrine. Although usually effective and safe, these drugs can redistribute blood flow in such a way as to compromise the splanchnic and renal circulation. Several mediators are thought to be responsible for producing postoperative shock, including bradykinin. For example, there is an inverse correlation between bradykinin concentrations and mean arterial pressure during CPB, suggesting that bradykinin is an important mediator in the decrease in SVR. We and others have shown that bradykinin induces vasodilation through its B2 receptor. In contract, B1 receptor stimulation does not cause vasodilation. As outlined under PRELIMINARY STUDIES, we have demonstrated that endogenous bradykinin contributes to protamine-related hypotension following CPB and that bradykinin receptor antagonism administered just prior to protamine attenuates this hypotensive response. In Specific Aim 2 we will test the hypothesis that bradykinin receptor antagonism modulate the hemodynamic changes observed during CPB.

Bradykinin receptor antagonism could reduce hyperfibrinolysis and CPB-associated blood loss. Inhibiting hyperfibrinolysis during CPB reduces blood loss and blood product requirements. On the other hand, modulating the hypofibrinolytic phase after CPB has the potential to reduce thrombotic complications. We and others have shown that bradykinin stimulates t-PA release from human forearm vasculature and the coronary circulation through a NO synthase-independent, and cyclooxygenase-independent pathway. As with vasodilation, bradykinin-stimulated t-PA release is mediated via the B2 receptor. Several groups have reported that bradykinin concentrations increase during CPB. We demonstrated a direct correlation between bradykinin and t-PA concentrations during CPB suggesting that bradykinin plays an important role in activating the fibrinolytic response during CPB. As outlined under PRELIMINARY STUDIES we have shown that HOE 140 (a B2 receptor antagonist) administered prior to CPB blunts the increase in D-dimer similar to e-aminocaproic acid. Thus, B2 receptor antagonism has the potential to reduce bradykinin-mediated fibrinolysis during CPB. In Specific Aim 2 we will test the hypothesis that bradykinin receptor antagonism modulate the fibrinolytic response observed during CPB.

Bradykinin receptor antagonism could reduce the inflammatory response to CPB. During CPB, exposure of blood to bioincompatible surfaces of the extracorporeal circuit, as well as tissue ischemia and reperfusion associated with the procedure, induce the activation of several major humoral pathways of inflammation. Bradykinin produces many of the characteristics of the inflammatory state, such as changes in local blood pressure, edema, and pain, resulting in vasodilation and increased microvessel permeability. Bradykinin activates NF-kB and upregulates interleukin(IL)-1b and TNFa-stimulated IL-8 production through the B2 receptor. In addition, bradykinin stimulates the release of IL-6 from a variety of cells. The growing knowledge of the biological role of kinins, in particular in inflammation, has fueled the development of potent and selective kinin receptor antagonist as potential therapeutics. For example, the bradykinin antagonist, deltibant (CP-0127) showed a significant improvement in the 28-day risk-adjusted survival of patients with gram-negative sepsis. In an animal model of intestinal ischemia-reperfusion injury, B2 receptor antagonism inhibited reperfusion induced increases in vascular permeability, neutrophil recruitment and expression of B1 receptor mRNA. The role of B2 receptor antagonist in myocardial ischemia-reperfusion injury is more controversial. Kumari et al demonstrated a protective effect of HOE 140 during in vivo ischemia-reperfusion injury, whereas in isolated rabbit heart studies, CP-0127 impaired recovery from acute coronary ischemia. This contradictory results may be the result of different antagonist used, differences in species sensitivity or different experimental protocols. The role of B1 receptor antagonist in inflammation is unclear. In contrast to the constitutively expressed bradykinin B2 receptor, bradykinin B1 receptor expression is upregulated following an inflammatory insult or ischemia-reperfusion injury. It appears that each kinin receptor subtype mediates different aspects of the inflammatory response. However, B1 receptor antagonism administered prior to CPB may be detrimental. For example, Siebeck et al demonstrated that B2 receptor blockade attenuates endotoxin-induced mortality in pigs, whereas additional B1 receptor blockade seemed to reverse these beneficial effects. Taken together, B2 receptor antagonism may decrease the acute inflammatory response whereas additional B1 receptor blockade may be harmful. These studies, and also the fact that aprotinin exerts part of its beneficial effects through a reduction in bradykinin concentrations, suggest the hypothesis that pharmacological strategies to block the bradykinin B2 receptor may be superior to reducing bradykinin concentrations in modulating the inflammatory response to CPB.

The RAS, KKS and inflammation. Activation of the RAS exerts proinflammatory effects. For example, Ang II activates the transcription factor nuclear factor (NF)-kB, which in turn regulates genes involved in cellular recruitment and the inflammatory cytokine cascade. Ang II induces the synthesis and secretion of the inflammatory interleukin (IL)-6. As mentioned above, bradykinin produces many of the characteristics of the inflammatory state and upregulates IL-1b and TNFa-stimulated IL-8 and stimulates the release of IL-6. Thus, both Ang II and bradykinin stimulates the release of IL-6. ACE inhibitor treatment is associated with a reduction in IL-6 response to CPB. In a randomized non-blinded study, Trevelyan and colleagues20 demonstrated that ACE inhibition produced a highly significant decrease of 51% in the release of IL-6 in patients identified as high producers of IL-6 by the -174 G/C polymorphism, whereas losartan had a similar but less marked effect. Potential mechanisms for this variation in IL-6 response between ACE inhibitors and angiotensin receptor blocker may be due to their differential effect on Ang II formation and bradykinin degradation. Furthermore, bradykinin-induced increases in IL-6 protein and total mRNA are inhibited by the selective B2 receptor antagonist HOE-140 but not by a selective B1 receptor antagonist. In Specific Aim 1 we will test the hypothesis that angiotensin-converting enzyme inhibitors and angiotensin II type 1 (AT1) receptor antagonist modulate the fibrinolytic and inflammatory response to CPB differently.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, 18 to 80 years of age, scheduled for elective CABG requiring CPB
2. For female subjects, the following conditions must be met:

postmenopausal for at least 1 year, or status-post surgical sterilization, or if of childbearing potential, utilizing adequate birth control and willing to undergo urine beta-hcg testing prior to drug treatment and on every study day

Exclusion Criteria:

1. Evidence of coagulopathy (INR greater than 1.7 without warfarin therapy)
2. Preoperative hematocrit less than 30%
3. Preoperative platelet count less than 100X109ml-1
4. GPIIb/IIIa antagonist within 48 hours of surgery
5. Emergency surgery
6. Impaired renal function (serum creatinine >1.6 mg/dl)
7. Pregnancy
8. Breast-feeding
9. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
10. History of alcohol or drug abuse
11. Treatment with any investigational drug in the 1 month preceding the study
12. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
13. Inability to comply with the protocol, e.g. uncooperative attitude and unlikelihood of completing the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mias Pretorius, MBChB, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - TN Valley Healthcare System, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Result] Balaguer JM, Yu C, Byrne JG, Ball SK, Petracek MR, Brown NJ, Pretorius M. Contribution of endogenous bradykinin to fibrinolysis, inflammation, and blood product transfusion following cardiac surgery: a randomized clinical trial. Clin Pharmacol Ther. 2013 Apr;93(4):326-34. doi: 10.1038/clpt.2012.249. Epub 2012 Dec 24. PMID 23361105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled by the research nurse at the time of the preoperative evaluation for surgery. All patients provided written informed consent. The study period was from June 2007 until June 2012.
Pre-assignment Details: One hundred and fifty patients consented to participate in the study. Of these patients, 13 were excluded,12 withdrew before randomization, 4 had their surgeries canceled, 3 had their surgery dates changed, and 3 patients did not proceed with the study for other reasons. The remaining 115 patients were randomly assigned to one of three groups.
Groups:
- Placebo Group: Normal saline (placebo) was started in the operating room after induction of anesthesia and before heparinization, continued throughout the bypass period, and discontinued at the end of surgery.
- Aminocaproic Acid Group: Aminocaproic acid (an antifibrinolytic drug) was started in the operating room after induction of anesthesia and before heparinization, continued throughout the bypass period, and discontinued at the end of surgery. Aminocaproic acid was given as an intravenous bolus of 100 mg/kg over one-half hour followed by an infusion of 30 mg/kg/hr.
- HOE 140 Group: HOE 140 (a bradykinin B2 receptor antagonist) was started in the operating room after induction of anesthesia and before heparinization, continued throughout the bypass period, and discontinued at the end of surgery. HOE 140 was given as an intravenous bolus of 22 µg/kg over one-half hour followed by an infusion of 18 µg/kg/hr.
Period: Overall Study
Arm/Group | Placebo Group | Aminocaproic Acid Group | HOE 140 Group
Started | 38 | 37 | 40
Completed | 38 | 37 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: Placebo was normal saline
- Aminocaproic Acid Group: Aminocaproic acid is an antifibrinolytic drug
- HOE 140 Group: Bradykinin B2 receptor antagonist
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Aminocaproic Acid Group | HOE 140 Group | Total
Number analyzed (Participants) | 38 | 37 | 40 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 23 | 24 | 72
  >=65 years | 13 | 14 | 16 | 43
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.8) | 58.5 (12.0) | 61.0 (12.8) | 59.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 18 | 48
  Male | 26 | 19 | 22 | 67
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 40 | 115

OUTCOME MEASURES:

1. Primary Outcome: Allogenic Blood Product Transfusion Risk
Description: Blood product transfusion during hospitalization that included packed red blood cells, plasma, platelets and cryoprecipitate.
Time Frame: Patients were followed for the duration of hospital stay, an average of 6 days
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Group | Aminocaproic Acid Group | HOE 140 Group
Number analyzed (Participants) | 38 | 37 | 40
percentage of participants
  Received any transfusion | 47.4 | 56.8 | 52.5
  Received packed red blood cells | 36.8 | 48.6 | 47.5
  Received plasma | 31.6 | 24.3 | 17.5
  Received platelets | 23.7 | 16.2 | 17.5
  Received cryoprecipitate | 10.5 | 2.7 | 5.0
Statistical Analysis 1: Comparison: Placebo Group vs Aminocaproic Acid Group vs HOE 140 Group; Test type: Superiority or Other; p = 0.72, Chi-squared — This P-value is for the main comparison of receiving any transfusion

2. Secondary Outcome: Units of Packed Red Blood Cells Transfused During Hospitalization
Description: Units of Packed Red Blood Cells Transfused
Time Frame: Patients were followed for the duration of hospital stay, an average of 6 days
Measure: Mean (Standard Error); unit: units
Arm/Group | Placebo Group | Aminocaproic Acid Group | HOE 140 Group
Number analyzed (Participants) | 38 | 37 | 40
units | 1.97 (0.61) | 1.41 (0.30) | 1.45 (0.34)
Statistical Analysis 1: Comparison: Placebo Group vs Aminocaproic Acid Group vs HOE 140 Group; Test type: Superiority or Other; p = 0.88, Kruskal-Wallis

3. Secondary Outcome: Units of Plasma Transfused During Hospitalization
Description: Units of plasma transfused
Time Frame: Patients were followed for the duration of hospital stay, an average of 6 days
Measure: Mean (Standard Error); unit: units
Arm/Group | Placebo Group | Aminocaproic Acid Group | HOE 140 Group
Number analyzed (Participants) | 38 | 37 | 40
units | 1.08 (0.37) | 0.68 (0.25) | 0.82 (0.36)
Statistical Analysis 1: Comparison: Placebo Group vs Aminocaproic Acid Group vs HOE 140 Group; Test type: Superiority or Other; p = 0.43, Kruskal-Wallis

4. Secondary Outcome: Inflammatory Response as Measured by Interleukin-6
Description: Interleukin-6 was measured at baseline, post-bypass and on postoperative day 1 and 2.
Time Frame: Patients were followed from the start of surgery until postoperative day 2
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo Group | Aminocaproic Acid Group | HOE 140 Group
Number analyzed (Participants) | 38 | 37 | 40
pg/ml
  Baseline | 4.98 (0.77) | 6.58 (1.50) | 4.80 (0.64)
  Post-bypass | 68.8 (17.49) | 64.65 (12.24) | 142.02 (85.28)
  Postoperative day 1 | 118.8 (19.15) | 161.91 (28.19) | 166.27 (49.44)
  Postoperative day 2 | 201.5 (95.29) | 122.88 (19.54) | 86.54 (15.84)
Statistical Analysis 1: Comparison: Placebo Group vs Aminocaproic Acid Group vs HOE 140 Group; The time course for Interleukin-6 concentrations were analyzed using mixed-effects models with fixed effects of drug treatment (placebo, aminocaproic acid, HOE 140) and time since randomization. We included a random subject effect and a first-order autoregressive process to account for the correlation in the response variable in the mixed-effects model; Test type: Superiority or Other; p = 0.92, Mixed Models Analysis — The P-value reflects the difference in Interleukin-6 concentrations among the 3 treatment groups over the course of the study (baseline, post-bypass, postoperative day 1 and 2)

5. Secondary Outcome: Fibrinolytic Response as Measured by D-dimer
Description: D-dimer concentrations were measured at baseline, 30min and 60min of bypass, post-bypass and postoperative day 1
Time Frame: Patients were followed from the start of surgery until postoperative day 1
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Placebo Group | Aminocaproic Acid Group | HOE 140 Group
Number analyzed (Participants) | 38 | 37 | 40
ng/ml
  Baseline | 95.5 (12.0) | 103.0 (18.8) | 88.1 (9.6)
  30min of bypass | 150.6 (17.5) | 131.9 (19.7) | 209.0 (49.4)
  60min of bypass | 287.6 (51.1) | 154.3 (24.7) | 363.3 (74.4)
  Post-bypass | 589.8 (104.5) | 168.9 (22.4) | 858.5 (182.5)
  Postoperative day 1 | 390.4 (73.2) | 269.5 (51.3) | 337.3 (36.4)
Statistical Analysis 1: Comparison: Placebo Group vs Aminocaproic Acid Group vs HOE 140 Group; The time course for D-dimer concentrations were analyzed using mixed-effects models with fixed effects of drug treatment (placebo, aminocaproic acid, HOE 140) and time since randomization. We included a random subject effect and a first-order autoregressive process to account for the correlation in the response variable in the mixed-effects model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value reflects the difference in D-dimer concentrations among the 3 treatment groups over the course of the study (baseline, 30min, 60min, post-bypass, and postoperative day 1)

ADVERSE EVENTS:
Time Frame: Hospitalization
Arm/Group | Placebo Group | Aminocaproic Acid Group | HOE 140 Group
Serious Adverse Events (participants affected / at risk) | 1/38 | 1/37 | 1/40
Other Adverse Events (participants affected / at risk) | 15/38 | 11/37 | 18/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=38) | Aminocaproic Acid Group (N=37) | HOE 140 Group (N=40)
Re-exploration for bleeding (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=38) | Aminocaproic Acid Group (N=37) | HOE 140 Group (N=40)
Acute kidney injury (Renal and urinary disorders) | 7 (7) | 4 (4) | 6 (6)
New onset postoperative atrial fibrillation (Cardiac disorders) | 5 (5) | 5 (5) | 9 (9)
Placement of permanent pacemaker (Cardiac disorders) | 2 (2) | 2 (2) | 3 (3)
Prolonged Mechanical Ventilation (>24 hours) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
This study was conducted in a population that predominantly underwent valve-only surgery. We cannot exclude the possibility that our results may have been different if we studied only coronary artery bypass graft surgery patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No